CLINICAL TRIAL: NCT07241988
Title: The Effect of Virtual Reality Glasses and White Noise on Pain, Anxiety, and Satisfaction During Peripheral Intravenous Catheterization in Adults: A Randomized Controlled Trial
Brief Title: Virtual Reality and White Noise During Peripheral IV Catheterization in Adults
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gizem Göktuna (Other)
Responsible Party: Sponsor-Investigator, Gizem Göktuna, Assistant Professor of Nursing, Dokuz Eylul University
Organization: Dokuz Eylul University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2025/31-10
Record Dates: First submitted 2025-11-17; First posted 2025-11-21 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Peripheral Intravenous Catheterization; Pain; Anxiety; Patient Satisfaction
Keywords: Virtual Reality; White Noise; Intravenous Catheterization; Pain; Anxiety
MeSH Terms: conditions — Pain; Anxiety Disorders; Patient Satisfaction

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Virtual Reality Group (Experimental): Participants in this group will wear virtual reality glasses displaying relaxing nature scenes during peripheral intravenous catheterization. The intervention will begin three minute before the procedure and continue until catheter insertion is completed.
  Interventions: Behavioral: Virtual Reality Glasses
- White Noise Group (Experimental): Participants in this group will listen to natural white noise (the sound of rain) through headphones during peripheral intravenous catheterization. The sound will begin three minutes before the procedure and continue until the catheterization is completed.
  Interventions: Behavioral: White Noise (Rain Sound)
- Control Group (No Intervention): Participants in this group will receive routine peripheral intravenous catheterization without any additional intervention.

INTERVENTIONS:
Behavioral: Virtual Reality Glasses — Participants in this group will wear virtual reality glasses displaying calming nature scenes accompanied by ambient sounds during peripheral intravenous catheterization. The intervention will begin three minutes before the procedure and continue until completion. This visual distraction technique is intended to reduce pain perception and anxiety levels and to increase patient satisfaction during the procedure.
  Other Names: VR Glasses
  Arms: Virtual Reality Group
Behavioral: White Noise (Rain Sound) — Participants will listen to natural white noise, specifically the sound of rain, through headphones during peripheral intravenous catheterization. The sound will begin three minutes before the procedure and continue until completion. This auditory distraction technique is intended to reduce pain perception and anxiety levels and to increase patient satisfaction during the procedure.
  Arms: White Noise Group

SUMMARY:
This randomized controlled study aims to examine the effects of using virtual reality glasses and white noise during peripheral intravenous catheterization on pain, anxiety, and satisfaction in adult patients. Participants will be randomly assigned to one of three groups: virtual reality, white noise, or control. Pain and anxiety levels will be assessed using standardized scales immediately after the procedure, and satisfaction will be evaluated following the intervention. The study aims to determine whether these non-pharmacological methods can reduce pain and anxiety and increase patient satisfaction during intravenous catheterization.

ELIGIBILITY:
Inclusion Criteria:

* No verbal, visual, auditory, or perceptual communication impairment
* Voluntary participation in the study
* Clinical requirement for peripheral intravenous catheterization
* No use of analgesic medication within the last 24 hours
* No diagnosed neurological or psychiatric disorder
* Ability to speak and understand Turkish
* Successful peripheral intravenous catheterization on the first attempt

Exclusion Criteria:

* Under 18 years of age
* Clinically unstable condition
* Individuals with psychiatric, mental, visual, or hearing impairments that prevent effective communication
* Individuals experiencing pain for any reason or using analgesic medication for pain management
* Individuals using anxiolytic or sedative medications
* Individuals who do not consent to participate in the study

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-10-11 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
ain intensity during peripheral intravenous catheterization | Immediately after peripheral intravenous catheterization
  Pain intensity will be measured using a Visual Analogue Scale (VAS) ranging from 0 (no pain) to 10 (worst possible pain) immediately after the procedure.

SECONDARY OUTCOMES:
Anxiety level during peripheral intravenous catheterization | Three minutes before and immediately after the peripheral intravenous catheterization
  Anxiety will be assessed using the State Anxiety Inventory-Short Form (STAIS-S). The scale measures temporary anxiety levels. Scores range from 5 to 20, with higher scores indicating higher (worse) anxiety. Measurements will be performed twice: three minutes before the intervention and immediately after the procedure is completed.
Patient satisfaction related to peripheral intravenous catheterization | Three minutes before and immediately after the peripheral intravenous catheterization
  Patient satisfaction will be assessed using a Visual Analogue Scale (VAS) ranging from 0 (not satisfied at all) to 10 (extremely satisfied). Measurements will be performed twice: three minutes before the procedure and immediately after the catheterization is completed. Higher scores indicate greater satisfaction.

CONTACTS AND LOCATIONS:
Locations (1):
- Dokuz Eylul University Hospital, İzmir, Balıkesir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) may be available from the principal investigator upon reasonable request.